CLINICAL TRIAL: NCT00003801
Title: Intergroup Rhabdomyosarcoma Study Group: Late Effects After Treatment for Rhabdomyosarcoma
Brief Title: Health-Related Outcomes in Patients Who Were Previously Treated for Rhabdomyosarcoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: Pediatric Oncology Group (Other); Children's Cancer Group (Other)
Purpose: Supportive Care
Other Study IDs: CDR0000066945; IRS-D9801; CCG-D9801; POG-D9801
Record Dates: First submitted 1999-11-01; First posted 2004-05-20 (Estimated); Last update posted 2009-08-20 (Estimated); Status verified 2000-02

CONDITIONS: Long-term Effects Secondary to Cancer Therapy in Children; Sarcoma
Keywords: long-term effects secondary to cancer therapy in children; previously treated childhood rhabdomyosarcoma
MeSH Terms: conditions — Sarcoma

INTERVENTIONS:
Procedure: management of therapy complications
Procedure: quality-of-life assessment

SUMMARY:
RATIONALE: Cancer treatment may have risks that affect health outcomes later. It is not yet known what health outcomes may be related to previous treatment for rhabdomyosarcoma.

PURPOSE: Study to determine health outcomes in patients who have survived 5 years after receiving treatment for rhabdomyosarcoma on the Intergroup Rhabdomyosarcoma Study Group protocols.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the frequency of self reported health related outcomes in patients with rhabdomyosarcoma who survived 5 years from diagnosis after treatment on Intergroup Rhabdomyosarcoma Study Group (IRSG) protocols I, II, III, and IV pilot. II. Determine the mortality of these patients and compare this mortality to the general population, especially in the third and fourth decades of life. III. Determine treatment specific risks of developing a second malignancy following treatment of rhabdomyosarcoma and the potential genetic influences (family history of cancer). IV. Determine the association between decreased fertility/offspring and dose, schedule, and total dose of alkylating agents (especially cyclophosphamide) received during treatment and with selected genitourinary and paratesticular primaries. V. Determine the effect of the dose and location of therapeutic radiation for primary head and neck cancer on achieved final height. VI. Determine the association of therapy with doxorubicin (dose and age when received) with cardiac and vascular events.

OUTLINE: Patients (or parent or surviving family member) complete the baseline questionnaire plus other questionnaires (offspring, family history, other topic specific). Medical data is also collected from past records.

PROJECTED ACCRUAL: Approximately 1600 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Prior registration on Intergroup Rhabdomyosarcoma Study Group Study IRS-I, IRS-II, IRS-III, IRS-IV pilot, IRS-V, or IRS-V pilot, or one of the protocols of IRS-V (D9501, D9502, D9602) AND Survived for 5 years after diagnosis (may be deceased now)

PATIENT CHARACTERISTICS: Age: 5 and over Performance status: Not specified Life expectancy: Not specified Hematopoietic: Not specified Hepatic: Not specified Renal: Not specified

PRIOR CONCURRENT THERAPY: See Disease Characteristics

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: William M. Crist, MD, Study Chair — University of Missouri-Columbia; Michael P. Link, MD, Study Chair — Stanford University; R. Beverly Raney, MD, Study Chair — M.D. Anderson Cancer Center